CLINICAL TRIAL: NCT00535002
Title: SCOR on Sex and Gender Factors Affecting Women's Health
Brief Title: The Effect of Yohimbine on Cocaine Cue Reactivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P50DA016511-1; P50DA016511 (NIH)
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-03

CONDITIONS: Cocaine Related Disorders
Keywords: Cocaine Addiction; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Yohimbine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cocaine Females, Yohimbine then Placebo (Other): Cocaine dependent females, received yohimbine day 1 and placebo day 2
  Interventions: Drug: Yohimbine; Drug: Placebo
- Cocaine Females, Placebo the Yohimbine (Other): Cocaine dependent females, received placebo day 1 and yohimbine day 2
  Interventions: Drug: Yohimbine; Drug: Placebo
- Cocaine Males, Yohimbine then Placebo (Other): Cocaine dependent males, received yohimbine day 1 and placebo day 2
  Interventions: Drug: Yohimbine; Drug: Placebo
- Cocaine Males, Placebo thenYohimbine (Other): Cocaine dependent males, received placebo day 1 and yohimbine day 2
  Interventions: Drug: Yohimbine; Drug: Placebo
- Control Females, Yohimbine then Placebo (Other): Non-dependent females, received yohimbine day 1 and placebo day 2
  Interventions: Drug: Yohimbine; Drug: Placebo
- Control Females, Placebo then Yohimbine (Other): Non-dependent females, received placebo day 1 and yohimbine day 2
  Interventions: Drug: Yohimbine; Drug: Placebo
- Control Males, Yohimbine then Placebo (Other): Non-dependent males, received yohimbine day 1 and placebo day 2
  Interventions: Drug: Yohimbine; Drug: Placebo
- Control Males, Placebo then Yohimbine (Other): Non-dependent males, received placebo day 1 and yohimbine day 2
  Interventions: Drug: Yohimbine; Drug: Placebo

INTERVENTIONS:
Drug: Yohimbine — Participants were pre-treated with either yohimbine or placebo.
Drug: Placebo

SUMMARY:
Stress and cues reminiscent of cocaine use promote craving and relapse in cocaine dependent individuals. In addition, there appears to be gender differences in determinants of relapse to drug use following abstinence in cocaine-dependent individuals. Therefore the purpose of the present study is to study the role of hormonal status on the response to cocaine-related cues with or without stress in cocaine-dependent women and men.

DETAILED DESCRIPTION:
Cocaine dependence is an insidious disease underscored by a strong propensity to relapse despite knowledge of the repercussions of continued drug-use. Stress and cocaine cues produce craving and ultimately relapse in cocaine dependent individuals. Pre-clinical research has demonstrated sex differences in response to cocaine-conditioned cues and cocaine-primed reinstatement, which correlates well with reduced plasma progesterone levels. Interestingly, this is consistent with a growing body of clinical literature indicating that progesterone may decrease the reinforcing properties of stimulants in women. Gender differences in the response to a social stressor and cocaine cues in cocaine-dependent individuals have been demonstrated in human laboratory studies, however, the interaction of stress and cues and the effect of hormonal status on response have not been explored. This study examines the role of hormonal status on the response to cocaine-related cues with or without a pharmacological stressor (yohimbine) in cocaine-dependent women and men. As a further integration of the research focus this study also explores the relationship between impulsivity and craving.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
* Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for a three-day period immediately prior to the CTRC admission. Nicotine dependence can affect HPA function (Baron et al., 1995) therefore it would be ideal to exclude subjects with nicotine use. Because of the high comorbidity of cocaine and nicotine dependence, this would seriously compromise the feasibility of recruitment. Individuals with alcohol dependence will be excluded. However because of the high comorbidity of alcohol use and cocaine dependence, individuals with alcohol abuse will be included. Also, due to the high comorbidity of cocaine and marijuana dependence, and limited evidence that marijuana use affects HPA function, subjects with marijuana dependence will be included.
* Subjects with ADHD will be included. Because ADHD is commonly characterized by impulsivity, ADHD severity ratings will be determined and controlled for in data analysis.
* Subjects must consent to random assignment.
* Subjects must consent to outpatient admission to the CTRC and two overnight admissions to the Medical University Hospital.

Exclusion Criteria:

* Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
* Women with premenstrual dysphoric disorder as this may impact on the response to the stress test procedure (Woods et al., 1994).
* Women receiving depot medroxyprogesterone acetate as a form of birth control.
* Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect physiological/subjective responses.
* Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect hormonal/neuroendocrine status.
* Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with subjective measurements.
* Subjects with current major depressive disorder or post-traumatic stress disorder as these disorders are associated with characteristic changes in stress response.
* Subjects with panic disorder, as yohimbine may precipitate panic attacks.
* Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents that interfere with hormonal measurements within one month of test session.
* Subjects taking any psychotropic medications,antidepressants, opiates or opiate antagonists because these may affect test response. Subjects taking SSRI's will be included.
* Subjects with any acute illness or fever. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
* Subjects who are obese (BMI>35) as this may interfere with hormonal status.
* Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for three days prior to the stress task procedure.
* Subjects meeting DSM-IV criteria for substance dependence (other than nicotine, alcohol, marijuana or cocaine as appropriate) within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen T Brady, M.D., Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina-GCRC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cocaine-dependent and control males and females between the ages of 18 and 65 were recruited between July 2008 and July 2012. Participants were primarily recruited through newspaper advertisements, and study procedures were conducted in the Clinical Neuroscience Division and Clinical and Translational Research Center of MUSC.
Pre-assignment Details: A total of 400 people consented to study participation; 171 met study inclusion criteria. 115 people completed study procedures, and the data of 112 subjects was included for analysis. Data from two participants were excluded from analysis because it was discovered later that they did not meet eligibility requirements.
Groups:
- Cocaine Females, Yohimbine Then Placebo: Cocaine-dependent females, Yohimbine then placebo
- Cocaine Males, Yohimbine Then Placebo: Cocaine-dependent males, Yohimbine then placebo
- Control Females, Yohimbine Then Placebo: Non-dependent females, Yohimbine then placebo
- Control Males, Yohimbine Then Placebo: Non-dependent males, Yohimbine then placebo
- Cocaine Females, Placebo Then Yohimbine: Cocaine females-dependent females, Placebo then yohimbine
- Cocaine Males, Placebo Then Yohimbine: Cocaine-dependent males, Placebo then Yohimbine
- Control Females, Placebo Then Yohimbine: Non-dependent females, placebo then yohimbine
- Control Males, Placebo Then Yohimbine: Non-dependent males, placebo then yohimbine
Period: Overall Study
Arm/Group | Cocaine Females, Yohimbine Then Placebo | Cocaine Males, Yohimbine Then Placebo | Control Females, Yohimbine Then Placebo | Control Males, Yohimbine Then Placebo | Cocaine Females, Placebo Then Yohimbine | Cocaine Males, Placebo Then Yohimbine | Control Females, Placebo Then Yohimbine | Control Males, Placebo Then Yohimbine
Started | 19 | 12 | 13 | 14 | 9 | 17 | 12 | 16
Completed | 19 | 12 | 13 | 14 | 9 | 17 | 12 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cocaine Females, Yohimbine Then Placebo: Cocaine-dependent females, received yohimbine day 1, placebo day 2
- Cocaine Females, Placebo Then Yohimbine: Cocaine-dependent females, received placebo day 1, yohimbine day 2
- Cocaine Males, Yohimbine Then Placebo: Cocaine-dependent males, received yohimbine day 1, placebo day 2
- Cocaine Males, Placebo Then Yohimbine: Cocaine-dependent males, received placebo day 1, yohimbine day 2
- Control Females, Yohimbine Then Placebo: non-dependent females, received yohimbine day and placebo day 2
- Control Females, Placebo Then Yohimbine: non-dependent females, received placebo day and yohimbine day 2
- Control Males, Yohimbine Then Placebo: non-dependent males, received yohimbine day and placebo day 2
- Control Males, Placebo Then Yohimbine: non-dependent males, received placebo day and yohimbine day 2
- Total: Total of all reporting groups
Arm/Group | Cocaine Females, Yohimbine Then Placebo | Cocaine Females, Placebo Then Yohimbine | Cocaine Males, Yohimbine Then Placebo | Cocaine Males, Placebo Then Yohimbine | Control Females, Yohimbine Then Placebo | Control Females, Placebo Then Yohimbine | Control Males, Yohimbine Then Placebo | Control Males, Placebo Then Yohimbine | Total
Number analyzed (Participants) | 19 | 9 | 12 | 17 | 13 | 12 | 14 | 16 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 9 | 12 | 17 | 13 | 12 | 14 | 16 | 112
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (10.1) | 37.8 (11.2) | 39.8 (10.9) | 38.7 (10.1) | 36.2 (13.2) | 32.1 (13.2) | 32.7 (13.3) | 32.3 (12.6) | 36.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 0 | 0 | 13 | 12 | 0 | 0 | 53
  Male | 0 | 0 | 12 | 17 | 0 | 0 | 14 | 16 | 59
Region of Enrollment [Number; unit: participants]
  United States | 19 | 9 | 12 | 17 | 13 | 12 | 14 | 16 | 112

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Craving
Description: Cocaine-dependent participants were pre-treated with either yohimbine or placebo provided subjective ratings of cocaine craving immediately following cocaine cue exposure.
  The scale used was the Within Sessions Ratings Scales (Childress AR, McLellan AT, O'Brien CP (1986) Conditioned responses in a methadone population. A comparison of laboratory, clinic, and natural settings. Journal of Substance Abuse Treatment 3:173-179.) Craving was rated on a scale of 0-10 with 0 being Not At All and 10 being Extremely.
Time Frame: Post cocaine cue exposure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cocaine Females Yohimbine: Cocaine-dependent females pre-treated with yohimbine
- Cocaine Females Placebo: Cocaine-dependent females pre-treated with placebo
- Cocaine Males Yohimbine: Cocaine-dependent males pre-treated with yohimbine
- Cocaine Males Placebo: Cocaine-dependent males pre-treated with placebo
Arm/Group | Cocaine Females Yohimbine | Cocaine Females Placebo | Cocaine Males Yohimbine | Cocaine Males Placebo | Control Females Yohimbine | Control Females Placebo | Control Males Yohimbine | Control Males Placebo
Number analyzed (Participants) | 28 | 28 | 30 | 30 | 25 | 25 | 30 | 30
units on a scale | 4.8 (3.6) | 3.4 (3.6) | 3.0 (2.9) | 2.7 (3.1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Groups:
- Cocaine Females: Cocaine-dependent females
- Cocaine Males: Cocaine-dependent males
- Control Females: Non-dependent females
- Control Males: Non-dependent males
Arm/Group | Cocaine Females | Cocaine Males | Control Females | Control Males
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30 | 0/25 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30 | 0/25 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes